CLINICAL TRIAL: NCT06350253
Title: Comparison Of Measured To Predicted Resting Metabolism
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Exercise Physiology, Ohio University
Other Study IDs: 22-X-187
Record Dates: First submitted 2024-03-29; First posted 2024-04-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-07

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- 18-24 years old: 18-24 years old
  Interventions: Diagnostic Test: Metabolic cart; Diagnostic Test: MedGem; Diagnostic Test: BIA
- 24-29 years old
  Interventions: Diagnostic Test: Metabolic cart; Diagnostic Test: MedGem; Diagnostic Test: BIA
- 30-39 years old
  Interventions: Diagnostic Test: Metabolic cart; Diagnostic Test: MedGem; Diagnostic Test: BIA
- 40-49 years old
  Interventions: Diagnostic Test: Metabolic cart; Diagnostic Test: MedGem; Diagnostic Test: BIA
- 50-60 years old
  Interventions: Diagnostic Test: Metabolic cart; Diagnostic Test: MedGem; Diagnostic Test: BIA

INTERVENTIONS:
Diagnostic Test: Metabolic cart — RMR measurement via metabolic cart
Diagnostic Test: MedGem — RMR measurement via MedGem
Diagnostic Test: BIA — RMR estimation from BIA analysis

SUMMARY:
The purpose of this study is to compare RMR values from the BIA, predicted equations, and indirect calorimetry.

DETAILED DESCRIPTION:
Resting metabolic rate (RMR) describes the number of calories a person utilizes while at rest. The gold standard measurement is via inspired and expired air using a metabolic cart. However, researchers have established estimation equations and the use of body composition analysis to predict RMR when a metabolic cart is unavailable. The accuracy of the predicted equations and whole-body bioelectrical impedance (BIA) machines that produce this data is unknown. Therefore, the purpose of this study is to compare RMR values from the BIA, predicted equations, and indirect calorimetry.

Aim 1: to compare measured RMR from indirect calorimetry to values provided by the InBody 770 BIA machine and to established gender and age-appropriate prediction equations.

Aim 2: to compare RMR measured from indirect calorimetry using a metabolic cart (Gold Standard) to the Medgem handheld indirect calorimeter (FDA approved device).

ELIGIBILITY:
Inclusion Criteria:

* Men & women, aged 18-60

Exclusion Criteria:

* Have any known or suspected metabolic diseases such as diabetes, thyroid disorder, or high cholesterol
* Have any known or suspected cardiovascular or pulmonary diseases such as hypertension
* Are currently on beta blockers, taking antihypertensives, or antidepressants
* Current smoker or quit less than a year ago
* Unwilling to provide finger stick and urine sample

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men & women, aged 18-60 in cohorts by age: 18-24, 24-29, 30-39, 40-49, and 50-60 years of age
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States